CLINICAL TRIAL: NCT02562586
Title: Is Drainage Necessary After Total Hip Replacement? A Randomized Controlled Trial
Brief Title: Is Drainage Necessary After Total Hip Replacement?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jose Ricardo Negreiros Vicente, Head of Hip Surgery Group, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEP 1055
Record Dates: First submitted 2015-08-17; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis, Hip
Keywords: Suction; Arthroplasty; Replacement; Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed Suction Drainage System (Active Comparator): Group 1: patients undergoing total hip replacement received a Closed Suction Drainage System for 24 hours after the surgical procedure
  Interventions: Device: Closed Suction Drainage System
- No Closed Suction Drainage System (No Intervention): Group 2: patients undergoing total hip replacement have not received a Closed Suction Drainage System after the surgical procedure

INTERVENTIONS:
Device: Closed Suction Drainage System — patients undergoing total hip replacement have received a closed suction drainage for 24 hours after the surgical procedure
  Arms: Closed Suction Drainage System

SUMMARY:
The goal of this study was to compare early results of Total Hip Replacement (THR) in 2 groups of patients: with and without closed suction drainage (CSD). Patients were followed for 3 months post operatively.

DETAILED DESCRIPTION:
After approval from the local ethical committee, patients undergoing Total Hip Replacement (THR) were included in this study. Patients with previous hip surgeries and coagulation disorders were not included. All patients were submitted to a non-cemented Total Hip Replacement (THR) through a Hardinge's approach. Before wound closure, a nurse opened an envelope containing the patient randomization: group 1 - with closed suction drainage (CSD) and group 2 - without closed suction drainage (CSD). In the group 1, a sub-fascial suction drain was used, and kept for 24 hours. Data collected included: mid-tigh circumference after 24 hours, blood transfusion, inflammatory blood markers C-Reactive Protein (CRP), Erythrocyte sedimentation rate (ESR) and leucogram, Harris Hip Score (HHS) after 3 months, and complications. Patients were followed for 3 months post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Primary Hip Arthroplasty
* Lateral Hardinge Approach
* Non-cemented Acetabular and Femoral Components
* Length of Skin Incision between 10 and 20 cm

Exclusion Criteria:

* Coagulative Disorders
* Previous Surgery in the same limb
* Age below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline red blood cells (RBC) | Pre-operative and 24 Hours Postoperative
  total RBC loss (mL) = [Uncompensated RBC loss (mL)] + [Compensated RBC loss (mL)] Uncompensated RBC loss (mL) = [Initial RBC (mL)] - [Final RBC (mL)] Compensated RBC loss (mL) = [Sum of RBCs received from the various sources of transfusion] Initial RBC (mL) = [Estimated blood volume (mL)] x [Initial Hct level (%)] at Day -1 Final RBC (mL) = [Estimated blood volume (mL)] x [Final Hct level (%)] at Day +3 Estimated blood volume (mL) = Women: [Body surface area (m2)] x 2430 Men: [Body surface area (m2)] x 2530 Body surface area (m2) = 0.0235 x [Height (cm)]0.42246 x [Weight (kg)]0.51456 Total blood loss at Hct level of 35% (mL) = [Total blood loss (mL)] / 0.35

SECONDARY OUTCOMES:
Mid thigh circumference (cm) | Pre-operative and 24 Hours Postoperative to 3 Months Postoperative
  Metric tape is placed midway between upper border of patella and superior anterior iliac spine
C-Reactive Protein (CRP) (mg/L) | 3,6 and 12 Weeks Postoperative
Erythrocyte sedimentation rate (ESR) (mm/h) | 3,6 and 12 Weeks Postoperative
Complications | during 3 months follow-up

OTHER OUTCOMES:
Visual Analogue Scale for Pain | Pre-operative and 24 Hours Postoperative
  Scores range from 0 (no pain) to 10 (worst possible pain)
Harris Hip Score Questionnaire | Pre-operative and 3 Months Postoperative
  <70 Poor 70 - 79 Fair 80-89 Good 90 -100 Excellent

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ricardo Negreiros Vicente, MD PhD, Principal Investigator — Hip Surgery Group Instituto Ortopedia e Traumatologia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo IOT-HCFMUSP
Locations (1):
- Instituto Ortopedia e Traumatologia do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo IOT-HCFMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Zhou XD, Li J, Xiong Y, Jiang LF, Li WJ, Wu LD. Do we really need closed-suction drainage in total hip arthroplasty? A meta-analysis. Int Orthop. 2013 Nov;37(11):2109-18. doi: 10.1007/s00264-013-2053-8. Epub 2013 Aug 28. PMID 23982636
- [Background] Gonzalez Della Valle A, Slullitel G, Vestri R, Comba F, Buttaro M, Piccaluga F. No need for routine closed suction drainage in elective arthroplasty of the hip: a prospective randomized trial in 104 operations. Acta Orthop Scand. 2004 Feb;75(1):30-3. doi: 10.1080/00016470410001708050. PMID 15022802
- [Background] Chen ZY, Gao Y, Chen W, Li X, Zhang YZ. Is wound drainage necessary in hip arthroplasty? A meta-analysis of randomized controlled trials. Eur J Orthop Surg Traumatol. 2014 Aug;24(6):939-46. doi: 10.1007/s00590-013-1284-0. Epub 2013 Aug 6. PMID 23917702
- [Background] Ovadia D, Luger E, Bickels J, Menachem A, Dekel S. Efficacy of closed wound drainage after total joint arthroplasty. A prospective randomized study. J Arthroplasty. 1997 Apr;12(3):317-21. doi: 10.1016/s0883-5403(97)90029-2. PMID 9113547
- [Background] Strahovnik A, Fokter SK, Kotnik M. Comparison of drainage techniques on prolonged serous drainage after total hip arthroplasty. J Arthroplasty. 2010 Feb;25(2):244-8. doi: 10.1016/j.arth.2008.08.014. Epub 2008 Dec 4. PMID 19056215
- [Background] Willett KM, Simmons CD, Bentley G. The effect of suction drains after total hip replacement. J Bone Joint Surg Br. 1988 Aug;70(4):607-10. doi: 10.1302/0301-620X.70B4.3403607.